CLINICAL TRIAL: NCT01959880
Title: CPG Styles Study: A Study of the Safety of the Contour Profile Gel Breast Implants in Subjects Who Are Undergoing Primary Breast Augmentation, Primary Breast Reconstruction or Revision
Brief Title: CPG Styles Study: A Study of the Safety of the Contour Profile Gel Breast Implants (CPG Styles Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110390SS-0313-2
Record Dates: First submitted 2013-09-25; First posted 2013-10-10 (Estimated); Results first posted 2016-11-11 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-09

CONDITIONS: Breast Augmentation; Breast Reconstruction; Breast Revision
Keywords: Breast Augmentation; Breast Reconstruction; Breast Revision; Silicone Gel; Contour Profile Gel; Siltex; CPG Styles
MeSH Terms: interventions — Breast Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Primary Augmentation (Other): The Augmentation cohort will include patients who have post-lactational mammary involution or wish general breast enlargement.
  Interventions: Device: The Contour Profile Gel (CPG) breast implants
- Primary Reconstruction (Other): The Reconstruction cohort will include patients with loss of breast due to mastectomy or with deformities secondary to disease, malignancy, trauma, and congenital deformity.
  Congenital deformities will include deformities of the breast itself as well as skeletal abnormalities reflected in breast deformity or asymmetry.
  Interventions: Device: The Contour Profile Gel (CPG) breast implants
- Revison Augmentation (Other): Patients in this cohort will have had previous breast augmentation with silicone or saline filled implants and are having a revision surgery to correct or improve the result of any previous breast augmentation surgery.
  Interventions: Device: The Contour Profile Gel (CPG) breast implants
- Revision Reconstruction (Other): Patients in this cohort will have had previous breast reconstruction with silicone or saline filled implants and are having a revision surgery to correct or improve the result of any previous breast reconstruction surgery.
  Interventions: Device: The Contour Profile Gel (CPG) breast implants

INTERVENTIONS:
Device: The Contour Profile Gel (CPG) breast implants — The CPG mammary prosthesis is a silicone elastomer mammary device with a textured surface. The Siltex® (textured) shell consists of a smooth shell bonded to an additional layer of silicone that has a textured pattern imprinted into its surface. The Siltex® shell is textured to provide a disruptive surface for collagen interface. The CPG implant contains a gel that is a more cohesive silicone gel than that used in other Mentor gel implants. The gel is made from the same materials as Mentor's standard gel. The contour shape of the CPG is designed to provide inferior projection with reduced superior fullness. The CPG mammary prosthesis contains raised orientation marks on the anterior and posterior of the implant which may help the physician ensure proper placement.
  The Contour Profile Gel is available in sizes 125cc - 690cc and 4 styles with various projection and height options in this study.

SUMMARY:
The CPG Styles Study is designed to demonstrate the safety of different styles of Mentor's Contour Profile Gel (CPG) breast implants in women who are undergoing primary augmentation, primary reconstruction, or revision. Safety information on the rate of capsular contracture, rupture and infection will be collected and used to determine device safety.

DETAILED DESCRIPTION:
Silicone gel-filled breast implants were introduced in the early sixties and were in wide-scale distribution by the time the Medical Device Amendments to the Food Drug and Cosmetic Act was passed in 1976. In 1983, gel-filled breast implants were designated as Class III devices requiring pre-market approval. In May 1990, the Food and Drug Administration (FDA) published a proposed request (515(b)) for Pre-market Approval Applications (PMA) and in April 1991 published the final request. This final publication put manufacturers of gel-filled breast implants on notice that for continued marketing of gel-filled breast implants, a PMA was due to FDA in 90 days from the final publication date.

A pre-market approval (PMA) for the Mentor gel-filled breast implants was filed with the FDA in July 1991. At the FDA General and Plastic Surgery Advisory Committee meeting in November 1991, the committee recommended the submission of additional information to establish the safety and effectiveness of gel-filled breast implants.

In January 1992, the FDA Commissioner announced a voluntary moratorium of the sale of gel-filled breast implants to allow the advisory panel time to assess additional information. In April 1992, the moratorium was lifted but only for reconstruction and revision subjects. Every subject implanted had to be part of an adjunct study, in addition to being offered participation in a registry of gel-filled breast implant subjects. In order to be implanted with gel-filled implants for augmentation, women had to be enrolled in an IDE clinical trial.

In September of 2000 the Core Gel study began, leading the way to the November 2006 FDA approval of MemoryGel breast implant.

The objective of the CPG Styles Study is to determine the safety of the different styles of Mentor's Contour Profile Gel (CPG) breast implants in women undergoing breast augmentation, reconstruction, or revision.

Throughout the duration of this study, patients are required to have follow-up visits at 10 weeks post-surgery and every year after surgery through the 10th year of study completion.

Total subject population: Up to 500 new subjects, plus up to 1500 subjects rolled over from the CPG Continued Access Study will continue the 10-year follow-up under this protocol.

On September 10th, 2014, Mentor received FDA approval for the CPG Styles 312, 322, 323, and 332. The study is now closed to new subject enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Subject is genetic female, 18 years of age or older
* A candidate for: Primary breast augmentation (general breast enlargement), Primary breast reconstruction (for trauma, loss of breast tissue due to mastectomy, malignancy, contralateral post-reconstruction symmetry, congenital deformity, including asymmetry), or Revision surgery (previous augmentation or reconstruction with silicone-filled or saline-filled implants)
* Signs the Informed Consent
* Agrees to return device to Mentor if explant necessary
* Agrees to comply with follow-up procedures, including returning for all follow-up visits

Exclusion Criteria:

* Subject is pregnant
* Has nursed a child within three months of study enrollment
* Been implanted with any silicone implant other than breast implants (e.g. silicone artificial joints or facial implants)
* Confirmed diagnosis of the following rheumatic diseases or syndromes: SLE, Sjogren's syndrome, scleroderma, polymyositis, or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondylarthropathies, any other inflammatory arthritis, fibromyalgia, or chronic fatigue syndrome
* Currently has a condition that could compromise or complicate wound healing (except reconstruction subjects)
* Subject in Augmentation cohort and has diagnosis of active cancer of any type. (Exception is low-grade non-metastasizing skin cancer)
* Infection or abscess anywhere in the body
* Demonstrates tissue characteristics which are clinically incompatible with implant (e.g. tissue damage resulting from radiation, inadequate tissue, or compromised vascularity)
* Possesses any condition, or is under treatment for any condition which, in the opinion of the investigator and/or consulting physicians(s), may constitute an unwarranted surgical risk
* Anatomic or physiologic abnormality which could lead to significant postoperative adverse events
* Demonstrates characteristics that are unrealistic/unreasonable with the risks involved with the surgical procedure
* Premalignant breast disease without a subcutaneous mastectomy
* Untreated or inappropriately treated breast malignancy, without mastectomy
* Are HIV positive
* Work for Mentor or the study doctor or are directly-related to anyone that works for Mentor or the study doctor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1891 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Canady, M.D., Study Director — Mentor Worldwide, LLC
Locations (1):
- Mentor Worldwide LLC, Santa Barbara, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Started | 1132 | 369 | 209 | 181
Completed | 0 (FDA granted approval for devices leading to early study completion. One subject reached 10 years.) | 0 (FDA granted approval for devices leading to early study completion. One subject reached 10 years.) | 1 (FDA granted approval for devices leading to early study completion. One subject reached 10 years.) | 0 (FDA granted approval for devices leading to early study completion. One subject reached 10 years.)
Not Completed | 1132 | 369 | 208 | 181
Not completed — Withdrawal by Subject | 11 | 13 | 8 | 7
Not completed — Death | 1 | 10 | 1 | 2
Not completed — Lost to Follow-up | 95 | 18 | 15 | 8
Not completed — Explantation w/o study device reimplant. | 22 | 17 | 5 | 12
Not completed — Study completed early-FDA approved | 1003 | 311 | 179 | 152

BASELINE CHARACTERISTICS:
Population: All subjects who signed informed consent and were implanted with MemoryGel breast implants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction | Total
Number analyzed (Participants) | 1132 | 369 | 209 | 181 | 1891
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (9.88) | 49.2 (10.58) | 46.7 (10.25) | 56.1 (9.37) | 40.7 (12.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1132 | 369 | 209 | 181 | 1891
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 58 | 5 | 2 | 3 | 68
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 15 | 14 | 0 | 4 | 33
  White | 986 | 334 | 192 | 162 | 1674
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 73 | 16 | 15 | 12 | 116
Region of Enrollment [Number; unit: participants]
  United States | 1132 | 369 | 209 | 181 | 1891

OUTCOME MEASURES:

1. Primary Outcome: 6-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Any Reoperation
Description: Time of occurrence calculated as the number of days from the date of the implant procedure to the onset date of the event. Patients were censored as of the date of their last office visit, the 120 month time point, or the date of explantation of all initial study devices, whichever was earliest.
Time Frame: 6 years
Population: All enrolled subjects are included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 1132 | 369 | 209 | 181
percentage of subjects | 8.3 [6.6 to 10.5] | 31.7 [25.5 to 39.1] | 13.8 [8.6 to 21.6] | 31.3 [23.8 to 40.4]

2. Primary Outcome: 6-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Baker III, IV Capsular Contracture
Description: Baker III was identified as "firm with visible distortion" and Baker IV was identified as "obvious spherical distortion". Time of occurrence calculated as the number of days from the date of the implant procedure to the onset date of the event. Patients were censored as of the date of their last office visit, the 120 month time point, or the date of explantation of all initial study devices, whichever was earliest.
Time Frame: 6 years
Population: All enrolled subjects are included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 1132 | 369 | 209 | 181
percentage of subjects | 1.5 [0.8 to 2.7] | 8.8 [5.3 to 14.4] | 1.6 [0.5 to 5.0] | 7.8 [3.6 to 16.6]

3. Primary Outcome: 6-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Infection
Description: as for outcome 1
Time Frame: 6 years
Population: All enrolled subjects are included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 1132 | 369 | 209 | 181
percentage of subjects | 1.0 [0.6 to 1.8] | 2.4 [1.2 to 4.8] | 1.0 [0.2 to 3.8] | 2.3 [0.9 to 6.0]

4. Primary Outcome: 6-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Explantation With or Without Replacement
Description: as for outcome 1
Time Frame: 6 years
Population: All enrolled subjects are included.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 1132 | 369 | 209 | 181
percentage of subjects | 5.0 [3.5 to 7.1] | 20.2 [14.6 to 27.5] | 8.6 [4.5 to 16.2] | 16.5 [10.9 to 24.6]

ADVERSE EVENTS:
Time Frame: Baseline (Surgery) to 6 Years
Description: Adverse events were collected as Complications in alignment with 2006 FDA Guidance. Consistent with this document, complications are not classified as serious or non-serious. Key safety endpoints are summarized under Outcome Measures. Complications are collected systematically using a pre-specified list of anticipated complications. No individual complications met the 5% threshold for reporting.
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Serious Adverse Events (participants affected / at risk) | 1/1132 | 10/369 | 1/209 | 2/181
Other Adverse Events (participants affected / at risk) | 0/1132 | 0/369 | 0/209 | 0/181
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Primary Augmentation (N=1132) | Primary Reconstruction (N=369) | Revison Augmentation (N=209) | Revision Reconstruction (N=181)
Death (General disorders) | 1 | 10 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator and his/her collaborators are free to publish the background, methods, and results of their own research without restraint. Prior review of any proposed manuscript or abstract will be provided to the sponsor to prevent premature disclosure of trade secrets or proprietary information. The review will occur 30 days prior to submission of manuscript or abstract for consideration of publication or to a conference. Sponsor reserves right to publish or present the overall study results.